CLINICAL TRIAL: NCT01217801
Title: Open-label Randomized, Two Way Crossover Bioequivalence Study to Compare Ondansetron Orally Dissolving FilmStrip 8mg With Zofran Orally Disintegrating Tablets 8 mg in 48 Healthy, Adult, Participants Under Fed Conditions.
Brief Title: Two Way Bioequivalence Study Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MonoSol Rx (Industry)
Responsible Party: Sponsor
Organization: Aquestive Therapeutics (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OND/CR/021/08-09/01906
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (ODFS) (Experimental): single dose of Ondansetron Orally Dissolving Filmstrip 8 mg
  Interventions: Drug: Ondansetron (ODFS)
- Zofran (ODT) (Active Comparator): Single dose of Zofran (Ondansetron) ODT Orally Disintegrating Tablets 8 mg
  Interventions: Drug: Ondansetron (ODT)

INTERVENTIONS:
Drug: Ondansetron (ODFS) — Ondansetron Orally Dissolving Filmstrip Ondansetron (ODFS)
  Other Names: Zuplenz
  Arms: Ondansetron (ODFS)
Drug: Ondansetron (ODT) — Ondansetron Orally Disintegrating Tablet Ondanestron (ODT)
  Other Names: Zofran
  Arms: Zofran (ODT)

SUMMARY:
The purpose of this study is to assess the single dose bioequivalence of Ondansetron ODFS 8mg with Zofran ODT® (Containing Ondansetron 8 mg) in healthy, male and female adult, human study participants under fed conditions.

The purpose is to monitor clinical status, adverse events, laboratory investigations and to assess relative safety and tolerance of ondansetron formulations under fed conditions.

DETAILED DESCRIPTION:
An open-label randomized, single oral dose, two way crossover bioequivalence study to compare ondansetron Orally Dissolving FilmStrip (ODFS) 8mg with Zofran Orally Disintegrating Tablets [ODT® (Containing Ondansetron 8 mg)] in 48 healthy, adult, human study participants under fed conditions. Volunteers who signed the consent form and showed their willingness to participate in the study were enrolled. Volunteers who satisfied the inclusion and exclusion criteria and found to be healthy on physical examination with laboratory investigation values within reference limits were considered eligible to be admitted into the study. Study participants were fasted for 10 hours prior to dosing in both periods. Dosing was conducted as per the randomization schedule in each period under fed conditions.A washout period of 7 days was observed between the two periods.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent.
* healthy adult within 18-45 years of age (inclusive).
* Body mass index of ≥ 18.5 kg/m2 and ≤ 25 kg/m2, with body weight not less than 50 kg.
* systolic blood pressure with upper limit of less than 140 mmHg and lower limit of more than or equal to 90 mm Hg.
* normal health as determined by medical history and physical examination performed within 15 days prior to the dosing of period 1.
* Normal ECG, chest X-ray and vital signs.
* If study volunteer is a female and is of child bearing potential practicing an acceptable method of birth control for the duration of the study.

Exclusion Criteria:

* The study participants were excluded based on the following criteria:

  * incapable of understanding the informed consent.
  * history of hypersensitivity or idiosyncratic reaction to study drug or any other related drug.
  * evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function
  * volunteers with a history of tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma .
  * smokes regularly more than ten cigarettes daily
  * taken over the counter or prescribed medications
  * history of any psychiatric illness, which may impair the ability to provide written, informed consent or full participation.
  * history of alcohol or substance abuse within the last 5 years.
  * clinically significant abnormal values of laboratory parameters.
  * positive urine screen for drugs of abuse at the time of admission check-in for each period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudershan Vishwanath, Study Director — Vimta VHS Research Centre
Locations (1):
- Vimta VHS Research Centre, Adyār, Chenni, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult study participants between 18-45 years (inclusive) of age who were willing to participate in the study by providing written informed consent
Groups:
- Ondansetron Orally Dissolving Filmstrip Then ODT: Ondansetron Orally Dissolving Filmstrip 8 mg then 7 days then Ondansetron Orally Disintegrating Tablet 8 mg measure AUC
- Ondansetron Orally Disintegrating Tablet Then OD Film: Ondansetron Orally Disintegrating Tablet AUC Ondansetron 8 mg then 7 days then Ondansetron Orally Disintegrating Film 8 mg measure AUC
Period: Period 1
Arm/Group | Ondansetron Orally Dissolving Filmstrip Then ODT | Ondansetron Orally Disintegrating Tablet Then OD Film
Started | 24 | 24
Completed | 23 | 22
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Ondansetron Orally Dissolving Filmstrip Then ODT | Ondansetron Orally Disintegrating Tablet Then OD Film
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study so the total number of participants is 48
Groups:
- Ondanestron Orally Dissolving Filmstrip: Ondanestron Orally Dissolving Filmstrip (8 mg) followed by a 7 day wash out and then administered Ondanestron Orally Disintegrating tablets (8 mg); AUCs for each period will be calculated.
- Ondanestron Orally Disintegrating Tablet: Ondanestron Orally Disintegrating Tablet (8 mg) followed by a 7 day wash out and then administered Ondanestron Orally Dissolving Filmstrip (8 mg); AUCs for each period will be calculated.
- Total: Total of all reporting groups
Arm/Group | Ondanestron Orally Dissolving Filmstrip | Ondanestron Orally Disintegrating Tablet | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.78 (5.8) | 26.78 (5.8) | 26.78 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  India | 48 | 48 | 48

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration
Description: Calculation of the AUC-Time Curve will be conducted to determine bio-equivalence.
Time Frame: Day 1 and Day 7
Population: All that completed a period
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Groups:
- Film: AUC film strip
- Tablet: tablet AUC
Arm/Group | Film | Tablet
Number analyzed (Participants) | 45 | 45
ng*hr/ml | 213.7 (47.8) | 225.9 (49.08)
Statistical Analysis 1: Comparison: Film vs Tablet; Linear mixed effect model, log transformed AUC, LSMeans for treatment Film and Tablet, the difference between the LSMeans and 90%CI calculated and transformed to geometric means, ratio estimates and 90%CI; Test type: Superiority or Other; p = 0.05, Regression, Linear; Hazard Ratio (HR) = 93.77, 90% CI 2-sided [89.15 to 98.63]

ADVERSE EVENTS:
Time Frame: study period Plus 30 days
Groups:
- Ondanestron Orally Dissolving Filmstrip: Ondanestron Orally Dissolving Filmstrip AUC
- Ondanestron Orally Disintegrating Tablet: Ondanestron Orally Disintegrating Tablet AUC
Arm/Group | Ondanestron Orally Dissolving Filmstrip | Ondanestron Orally Disintegrating Tablet
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 4/48 | 0/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ondanestron Orally Dissolving Filmstrip (N=48) | Ondanestron Orally Disintegrating Tablet (N=48)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) — film
URTI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — post study end received both dose forms
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — film

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes